CLINICAL TRIAL: NCT04602533
Title: A Phase II Randomized Study to Evaluate the Efficacy and Safety of Cisplatin or Carboplatin / Etoposide and Concomitant Radiotherapy Combined With Durvalumab Followed by Maintenance Therapy With Durvalumab Versus Cisplatin or Carboplatin / Etoposide and Concomitant Radiotherapy in Patients With Limited Disease Small Cell Lung Cancer
Brief Title: Efficacy and Safety of Standard of Care Plus Durvalumab in Patients With Limited Disease Small Cell Lung Cancer (DOLPHIN)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Hopp (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Michael Hopp, Head of Interdisciplinary Center for Clinical Studies (IZKS), Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dolphin; 2020-001050-22 (EudraCT Number)
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Small Cell Lung Cancer Limited Stage
Keywords: LD-SCLC; lung cancer; durvalumab
MeSH Terms: conditions — Lung Neoplasms | interventions — durvalumab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Durvalumab (Experimental): Induction phase: Durvalumab (1500 mg once every 3 weeks) for 4-6 cycles in combination with standard of care (Radiochemotherapy)
  Maintenance phase: Durvalumab (1500 mg once every 4 weeks) until PD or unacceptable toxicities.
  Interventions: Drug: Durvalumab
- standard of care (Other): Induction phase: Radiochemotherapy according to guideline
  Maintenance: Standard of care
  Interventions: Drug: standard of care

INTERVENTIONS:
Drug: Durvalumab — Induction phase: Durvalumab (1500 mg once every 3 weeks) for 4-6 cycles in combination with standard of care (Radiochemotherapy) Maintenance phase: Durvalumab (1500 mg once every 4 weeks) until PD or unacceptable toxicities.
  Other Names: IMFINZI®
  Arms: Durvalumab
Drug: standard of care — Radiochemotherapy: Cisplatin (75 mg/m² (BSA) D1#) or alternatively Carboplatin (AUC 5 D1) and Etoposide (100 mg/m² (BSA) D1-3) once every 3 weeks for 4-6 cycles and concomitant Radiotherapy (60±6 Gy, 1.8-2 Gy/d or 45±1.5 Gy (1.5 Gy per fraction twice daily, with 4 hours or more between fractions) with start at latest at beginning of cycle 3, ideally during cycle 1) followed by prophylactic cranial irradiation (PCI, if clinically indicated and according to local standard at any time after completion of radio-chemotherapy))
  A simultaneous administration of platinum-based chemotherapy (preferred Cisplatin) and radiotherapy for at least 2 cycles should be performed.
  Arms: standard of care

SUMMARY:
Combination of concomitant Radio-Chemotherapy showed a significant improvement (Takada) of OS and PFS in limited disease SCLC patients. This clinical trial is a prospective, multicenter, randomized, open-label, parallel group phase II investigator initiated trial (ITT) to evaluate the efficacy and safety of Durvalumab in combination with Cisplatin/Etoposide/Radiotherapy in patients with limited disease small-cell lung cancer (SCLC).

DETAILED DESCRIPTION:
The trial is subdivided in a safety run-in phase and a randomized part with the induction phase (Radiochemotherapy ± Durvalumab and including prophylactic cranial irradiation (PCI; if clinically indicated and according to local standard)) followed by the maintenance phase. The trial starts with the safety run-in phase of 6 patients in Durvalumab group. After the completion of the first cycle of all 6 patients a safety interim analysis will be performed. Study should be discontinued if ≥ 2 out of 6 patients within safety run-in phase (first cycle):

* show more than 2 AEs CTCAE grade ≥3 related to study drug Durvalumab
* or develop pneumonitis (CTCAE grade ≥2)
* or drop out, Otherwise, the trial can continue with randomization. Eligible patients will be randomized to Durvalumab group or standard of care group 2:1.

The safety interim analysis was performed in Q4 2021. The independent DMC has recommended the continuation of the trial.

Induction phase:

Durvalumab group: Cisplatin (75 mg/m² (BSA) D1#) or alternatively Carboplatin (AUC 5 D1) and Etoposide (100 mg/m² (BSA) D1-3) once every 3 weeks for 4-6 cycles and concomitant Radiotherapy (60±6 Gy, 1.8-2 Gy/d or 45±1.5 Gy (1.5 Gy per fraction twice daily, with 4 hours or more between fractions) with start at latest at beginning of cycle 3, ideally during cycle 1) and additional Durvalumab (1500 mg once every 3 weeks) for 4-6 cycles according to randomization followed by prophylactic cranial irradiation (PCI, if clinically indicated and according to local standard at any time after completion of radio-chemotherapy))

Control group: Cisplatin (75 mg/m² (BSA) D1#) or alternatively Carboplatin (AUC 5 D1) and Etoposide (100 mg/m² (BSA) D1-3) once every 3 weeks for 4-6 cycles and concomitant Radiotherapy (60±6 Gy, 1.8-2 Gy/d or 45±1.5 Gy (1.5 Gy per fraction twice daily, with 4 hours or more between fractions with start at latest at beginning of cycle 3, ideally during cycle 1) followed by prophylactic cranial irradiation (PCI, if clinically indicated and according to local standard at any time after completion of radio-chemotherapy)

# Due to the potential toxicity of Cisplatin 75 mg/m² D1, a Cisplatin split dose with 40 mg/m² on D1 and D8 is alternatively allowed. A switch from Cisplatin to Carboplatin AUC 5 D1 (due to new contraindication to Cisplatin) or split dose Carboplatin (AUC 2.5 D1 and D8) is also allowed. In case of initial contraindication to Cisplatin (i.e. renal dysfuction) at baseline, treatment can be started with Carboplatin once every 3 weeks (q21) AUC 5 D1, or split dose AUC 2.5 D1 and D8. A simultaneous administration of platinum-based chemotherapy (preferred Cisplatin) and radiotherapy for at least 2 cycles should be performed.

Maintenance phase:

In Durvalumab group patients will be treated with Durvalumab once every 4 weeks until disease progression (radiologic or clinical progression) or unacceptable toxicities, if patients show at least stable disease after induction phase. Patients with PD after induction phase will have EoT visit and will be followed up until death.

Patients in control group will have EoT visit and will receive standard of care treatment until PD and thereafter will be followed up until death.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent of the subject must be available before start of any specific trial procedures
* Male or female ≥ 18 years
* Histological confirmed limited disease small cell lung cancer (stage 2 and 3; T1a-4, N1-3, M0 according UICC8 criteria; if primarius is not eligible as RECIST1.1 target lesion (in cases with T1a and T1b) at least one lymph node must meet RECIST1.1 criteria for target lesion (≥15 mm short axis))
* Availability of tumor tissue or fresh tumor material for translational research by central lab testing
* ECOG PS 0 - 1
* At least one measurable lesion according RECIST 1.1
* Body weight > 30 kg
* Adequate normal organ function

  1. Hemoglobin ≥ 9.0 g/dL
  2. Absolute neutrophil count (ANC) ≥ 1.5 x109/L
  3. Platelet count ≥ 100 x109/L
  4. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal
  5. Serum Bilirubin ≤ 1.5 x institutional upper limit of normal
  6. Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min for Carboplatin, ≥ 60 mL/min for Cisplatin, calculated by the Cockcroft-Gault formula
* Life expectancy of at least 12 weeks in the discretion of the investigator
* Ability of subject to understand nature, importance and individual consequences of clinical trial

Exclusion Criteria:

* Extensive disease small cell lung cancer (Tx, Nx, M1; stage IV)
* Major surgical process within 28 day prior first dose of IMP and/or Radiochemotherapy
* History of allogenic organ transplantation
* Active or prior documented autoimmune or inflammatory disorder (including inflammatory bowel disease [e.g. colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome or Wegener syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.). The following are exceptions to this criterion:

  1. Patients with vitiligo or alopecia
  2. Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement
  3. Patients with any chronic skin condition that not required systemic therapy
  4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  5. Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness (i.e. active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, interstitial lung disease, serious chronic gastrointestinal conditions (i.e. diarrhea), psychiatric illness)
* History of another primary malignancy in the last 5 years, except adequately treated nonmelanoma skin cancer, adequately treated carcinoma in situ (without evidence of disease)
* History of leptomeningeal carcinomatosis, or brain metastases
* Known HIV positive and/or active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Current or prior use of immunosuppressive medication within 14 days before the first dose.The following are exceptions to this criterion:

  1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  2. Systemic corticosteroids at physiologic doses not exceeding 10 mg/day of prednisone or its equivalent
  3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IMP
* Participation in another clinical trial with an investigational product within the last 30 days (unless during follow-up period of an interventional study)
* Known hypersensitivity to one of the ingredients
* Medical or psychological conditions that would jeopardize an adequate and orderly completion of the trial
* Pregnancy, lactation and contraception

  1. Women who are pregnant, nursing or who plan to become pregnant while in the trial
  2. Women of child-bearing potential (WOCBP) and men who are able to father a child, unwilling to be abstinent or use highly effective methods of birth control that result in a low failure rate of less than 1% per year when used consistently and correctly beginning at informed consent, for the duration of drug treatment and for the drug out washout period (90 days after last dose of Durvalumab and/or 6 months after last dose of cisplatin/carboplatin and etoposide).
* Patients who are legally institutionalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 18 months
  Progression-free survival (PFS) after 18 months according to iRECIST

SECONDARY OUTCOMES:
Progression-free survival (PSF) after other assessments | 12 months
  Time between first application of trial medication to date of disease progression or death due to any cause
Overall survival (OS) | 18 months
  Time between first application of trial medication to date of death due to any cause
Overall response rate (ORR) | 18 months
  Complete Response or Partial Response according to iRECIST
Disease control rate (DCR) | 18 months
  Complete Response, Partial Response or Stable Disease according to iRECIST
Quality of Life Questionnaire - Cancer 30 (QLQ-C30) | 18 months
  Symptom control assessed by patient-reported quality of life (QoL) with QLQ-C30. The score ranges from 0 to 100. The higher the score the better the outcome.
Quality of Life Questionnaire - Lung Cancer 13 (QLQ-LC13) | 18 months
  Symptom control assessed by patient-reported quality of life (QoL) with QLQ-LC13. The scores ranges from 0 to 100. The higher the score the better the outcome.
EuroQol five dimension scale (EQ-5D) | 18 months
  Symptom control assessed by patient-reported quality of life (QoL) with EQ-5D. The score consists of 5 items on a three step scale and a VAS scale ranging from 0 to 100. The lower the score on the three step scales the better the outcome and the higher the score on the VAS scale the better the outcome.
Adverse Events | 18 months
  Treatment emergent adverse events during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wehler, Prof, Principal Investigator — Universitätsklinikum Gießen Marburg
Locations (16):
- Germany (16):
  - Klinik Löwenstein gGmbH, Löwenstein, Baden-Würtemberg
  - Klinikverbund Allgäu gGmbH, Immenstadt im Allgäu, Bavaria
  - Asklepios Fachkliniken Muenchen Gauting, München Gauting, Bavaria
  - Klinikum Ernst von Bergmann, Potsdam, Brandenburg
  - Universitätsklinikum Gießen Marburg, Giessen, Hesse
  - Klinikum Kassel GmbH-Klinik für Onkologie und Hämatologie, Kassel, Hesse
  - Sana-Klinikum Offenbach, Offenbach, Hesse
  - Universitätsmedizin Rostock, Rostock, Mecklenburg-Vorpommern
  - Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia
  - Lungenklinik Köln-Merheim, Cologne, North Rhine-Westphalia
  - KEM GmbH, Essen, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Lungenklinik Hemer, Hemer, North Rhine-Westphalia
  - Johannes Wesling Klinikum Minden, Minden, North Rhine-Westphalia
  - Helios Kliniken Erfurt, Erfurt, Thuringia
  - Asklepios Klinikum Hamburg, Hamburg

IPD SHARING:
Plan to Share IPD: No